CLINICAL TRIAL: NCT04998539
Title: Effect of Travel Direction, Body Position and Technique on the Ease of a Caregiver Getting an Occupied Wheelchair Over a Soft Surface: a Randomized Crossover Trial
Brief Title: Effect of Travel Direction, Body Position and Technique on the Ease of Getting an Occupied Wheelchair Over a Soft Surface
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Principal Investigator, Lee Kirby, Principal Investigator, Nova Scotia Health Authority
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: WSP-2021PP; 1027105 (Other: Nova Scotia Health REB)
Record Dates: First submitted 2021-07-16; First posted 2021-08-10 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Wheelchairs

STUDY DESIGN:
Intervention Model Description: This study consists of a randomized crossover trial with within-participant comparisons.
Who Masked: Participant
Masking Description: The participants will be blinded to the expected differences among the test conditions and asked not to discuss their experiences with other potential participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Upright wheelchair forward and occupant upright (Experimental): Participant will push an upright wheelchair forward over a 5 m soft surface with the wheelchair occupant in the upright body position. The participant will perform the task once.
  Interventions: Other: Wheelchair forward direction; Other: Upright technique; Other: Wheelchair occupant upright body position
- Upright wheelchair backward and occupant upright (Experimental): Participant will pull an upright wheelchair backwards over a 5 m soft surface with the wheelchair occupant in the upright body position. The participant will perform the task once.
  Interventions: Other: Wheelchair backward direction; Other: Upright technique; Other: Wheelchair occupant upright body position
- Wheelie wheelchair forward and occupant upright (Experimental): Participant will push a wheelchair using the wheelie technique forward over a 5 m soft surface with the wheelchair occupant in the upright body position.The participant will perform the task once.
  Interventions: Other: Wheelchair forward direction; Other: Wheelie technique; Other: Wheelchair occupant upright body position
- Wheelie wheelchair backward and occupant upright (Experimental): Participant will pull a wheelchair using the wheelie technique backwards over a 5 m soft surface with the wheelchair occupant in the upright body position.The participant will perform the task once.
  Interventions: Other: Wheelchair backward direction; Other: Wheelie technique; Other: Wheelchair occupant upright body position

INTERVENTIONS:
Other: Wheelchair forward direction — Participants will move the wheelchair over 5 meters of a soft surface (gym mats) in the forward direction. Participants will push the wheelchair when moving forward.
  Arms: Upright wheelchair forward and occupant upright; Wheelie wheelchair forward and occupant upright
Other: Wheelchair backward direction — Participants will move the wheelchair over 5 meters of a soft surface (gym mats) in the backward direction. Participants will pull the wheelchair when moving backwards.
  Arms: Upright wheelchair backward and occupant upright; Wheelie wheelchair backward and occupant upright
Other: Upright technique — Participants will move the wheelchair across the 5 m soft surface using the upright technique. The upright technique involves the wheelchair being moved with all 4 wheels on the ground.
  Arms: Upright wheelchair backward and occupant upright; Upright wheelchair forward and occupant upright
Other: Wheelie technique — Participants will move the wheelchair across the 5 m soft surface using the wheelie technique. The wheelie technique involves the wheelchair being tipped backward and balanced on the rear wheels. Participant wheelchair occupants will always be upright when being moved using the wheelie technique.
  Arms: Wheelie wheelchair backward and occupant upright; Wheelie wheelchair forward and occupant upright
Other: Wheelchair occupant upright body position — The participant occupying the wheelchair (wheelchair occupant) will be seated with a body position that is upright (back is leaning against the wheelchair back rest and arms on wheelchair arm rests) while the wheelchair is being moved.

SUMMARY:
Wheelchair skills training is an important step in the wheelchair provision process. Caregivers play an important role in the lives of wheelchair users but very little is known about wheelchair skills training for caregivers. The goal of the study is to understand the effect of wheelchair travel direction, wheelchair occupant body position and technique used by caregivers on the ease of getting an occupied wheelchair over a soft surface.

DETAILED DESCRIPTION:
Able bodied participants will be used to simulate caregivers and wheelchair occupants. Participants simulating caregivers will be asked to move the occupied wheelchair over a 5 m soft surface. Participants will be randomly assigned a direction to move the wheelchair (forward or backwards), wheelchair occupant body position (upright or leaning forward) and technique in moving the wheelchair (upright with all 4 wheels on ground or in a wheelie position with the wheelchair tipped backwards and balanced on the rear wheels). The ease of getting the occupied wheelchair over the soft surface will be evaluated by the amount of time taken to complete the task, how well the participant completed the task and the ease of performing the task as evaluated by the participant.

ELIGIBILITY:
Inclusion Criteria:

* able to communicate in English,
* alert, cooperative, and competent to provide informed consent,
* willing to participate (as evidenced by attending the single data-collection session), and
* have no physical impairments that would prevent their being able to push and pull a wheelchair over a soft surface

Exclusion Criteria:

* have unstable medical conditions that might make the handling of a manual wheelchair dangerous, or emotional problems that might make participation unsafe or unpleasant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Time taken to perform task | through study completion , an average of 1 hour
  The amount of time in seconds taken to perform the task and move the occupied wheelchair across 5 meters of soft surface (gym mats).

SECONDARY OUTCOMES:
Ability to perform task | through study completion , an average of 1 hour
  The ability of the participant to perform the task of moving the occupied wheelchair across the 5 meter soft surface. Participant will be scored using an ordinal scale from 0 to 3 (0 = fail, distance completed < 2.5 m and /or time taken more than 20 seconds, 1=partial pass with distance completed between 2.5 m and 4.9 m and time less than or equal to 20 seconds, 2 = pass with completion of the 5 m distance and time taken between 11 and 20 seconds, and advanced pass = 3 with completion of the 5 m distance and time taken being less than or equal to 10 seconds).
Ease of performing the task | through study completion , an average of 1 hour
  Participant self-reported ease of performing the task of moving the occupied wheelchair over a 5 meter soft surface. A five-point Likert scale with 4 = "very easy", 3 = "somewhat easy", 2 = "neither easy nor difficult", 1 = "somewhat difficult" and 0 = "very difficult".

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Rehabilitation and Arthritis Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Kirby RL, Parker K, Poon E, Smith C, Osmond D, Ladouceur M, Haworth VS, Theriault CJ, Sandila N. Effect of travel direction and wheelchair position on the ease of a caregiver getting an occupied wheelchair across a soft surface: a randomized crossover trial. Disabil Rehabil Assist Technol. 2024 May;19(4):1298-1306. doi: 10.1080/17483107.2023.2170476. Epub 2023 Jan 25. PMID 36695416